CLINICAL TRIAL: NCT00734474
Title: A Phase 2/3, Placebo-Controlled, Efficacy and Safety Study of Once-Weekly, Subcutaneous LY2189265 Compared to Sitagliptin in Patients With Type 2 Diabetes Mellitus on Metformin
Brief Title: A Study of LY2189265 Compared to Sitagliptin in Participants With Type 2 Diabetes Mellitus on Metformin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: United BioSource, LLC (Industry); Tessella Inc. (Industry); Berry Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11422; H9X-MC-GBCF (Other: Eli Lilly and Company); CTRI/2009/091/000969 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2015-01-28 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 3.0 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 3.0 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- 2.0 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 2.0 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- 1.5 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- 1.0 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 1.0 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- 0.75 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- 0.5 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 0.5 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- 0.25 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 0.25 milligrams (mg), subcutaneous (SC) injection, once weekly for up to 104 weeks
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
  Interventions: Drug: LY2189265; Drug: Placebo tablet; Drug: Metformin
- Sitagliptin (Active Comparator): Sitagliptin: 100-milligrams (mg) tablet, administered orally, once daily for 104 weeks
  Placebo: solution, subcutaneous (SC) injection, once weekly for 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
  Interventions: Drug: Sitagliptin; Drug: Placebo solution; Drug: Metformin
- Placebo/Sitagliptin (Baseline Through 104 Weeks) (Placebo Comparator): Placebo: solution, subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 26 weeks
  Sitagliptin: after 26 weeks, 100-milligrams (mg) tablet, administered orally, once daily for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
  Interventions: Drug: Placebo solution; Drug: Placebo tablet; Drug: Metformin

INTERVENTIONS:
Drug: LY2189265
  Other Names: Dulaglutide; Trulicity
  Arms: 0.25 mg LY2189265; 0.5 mg LY2189265; 0.75 mg LY2189265; 1.0 mg LY2189265; 1.5 mg LY2189265; 2.0 mg LY2189265; 3.0 mg LY2189265
Drug: Sitagliptin
  Arms: Sitagliptin
Drug: Placebo solution
  Arms: Placebo/Sitagliptin (Baseline Through 104 Weeks); Sitagliptin
Drug: Placebo tablet
  Arms: 0.25 mg LY2189265; 0.5 mg LY2189265; 0.75 mg LY2189265; 1.0 mg LY2189265; 1.5 mg LY2189265; 2.0 mg LY2189265; 3.0 mg LY2189265; Placebo/Sitagliptin (Baseline Through 104 Weeks)
Drug: Metformin

SUMMARY:
This is an adaptive dose finding study and a Phase 3 efficacy study to evaluate the effects of once weekly injection of LY2189265 compared to Sitagliptin on glucose by measuring glycosylated hemoglobin (HbA1c) change from baseline after 52 weeks in participants with type 2 diabetes mellitus on Metformin.

DETAILED DESCRIPTION:
This is a double blind study designed to select 1 or 2 LY2189265 doses for evaluation in Phase 3 studies (dose-finding portion) and to evaluate efficacy and safety of selected doses of LY2189265 in comparison to Sitagliptin (100 milligrams) up to 104 weeks and Placebo up to 26 weeks in participants with type 2 diabetes mellitus on Metformin (confirmatory, Phase 3 portion). The primary objective is to show non-inferiority of the higher LY2189265 dose (if 2 doses are selected) to Sitagliptin with respect to change in glycosylated hemoglobin (HbA1c) at 52 weeks. The final endpoint is 104 weeks.

Participants are randomized to receive Placebo, Sitagliptin, or 1 of 7 initial LY2189265 doses until a dose decision is made based on quantitative analysis of the benefits and risks of each LY2189265 dose. A clinical utility index (CUI) that applies predicted values for change from baseline in HbA1c at 12 months and change from baseline in weight, diastolic blood pressure, and pulse rate at 6 months for each LY2189265 dose will be used toward this end. After the dose decision, participants in the selected LY2189265 arms and the comparator arms (Sitagliptin and Placebo/Sitagliptin arms) will continue the study, and additional participants will be randomized to the selected and comparator arms. Regardless of the timing of randomization relative to the dose decision point, all participants in the selected and comparator arms are planned to receive treatment for 104 weeks; participants in the Placebo/Sitagliptin arm will receive Placebo treatment for 26 weeks followed by Sitagliptin 100 mg for 78 weeks for blinding purposes only, and participants in the selected and Sitagliptin arms will receive the same treatment for 104 weeks. All participants will remain blinded to their study treatment throughout the study. Participants in the non-selected arms will discontinue from the study after the dose decision

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type 2, for at least 6 months
* Treatment regimens: diet and exercise, metformin as monotherapy or in combination with another oral antihyperglycemic medication (OAM), or another OAM as monotherapy. Must be able to tolerate metformin at a dose of at least 1500 milligrams (mg) daily for 6 weeks prior to randomization.
* Glycosylated hemoglobin (HbA1c) value of ≥7.0% to ≤9.5%, except participants on diet and exercise therapy who must have had HbA1c value of >8.0% to ≤9.5%
* Body mass index (BMI) between 25 and 40 kilograms per meter squared (kg/m^2), inclusive
* Stable weight for 3 months prior to screening
* Females of childbearing potential must test negative for pregnancy and agree to use a reliable birth control method

Exclusion Criteria:

* Diabetes mellitus, type 1
* Use of a glucagon-like peptide-1 (GLP-1) analog (for example, exenatide) within 6 months prior to screening or are being treated with insulin
* Gastric emptying abnormality, history of bariatric surgery, or chronic use of drugs that affect gastrointestinal motility
* Use of medications to promote weight loss
* Clinically-relevant cardiovascular event within 6 months prior to screening
* Poorly controlled hypertension
* Electrocardiogram (ECG) reading considered outside the normal limits or indicating cardiac disease
* Liver disease, hepatitis, chronic pancreatitis, idiopathic acute pancreatitis, or alanine transaminase (ALT) levels >3.0 times the upper limit of normal
* Serum creatinine ≥1.5 milligrams per deciliter (mg/dL) or a creatinine clearance <60 milliliters per minute (mL/minute)
* Uncontrolled diabetes, defined as >2 episodes of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to study entry.
* Uncontrolled endocrine or autoimmune abnormality
* History of a transplanted organ
* Chronic use of systemic glucocorticoid therapy
* Active or untreated malignancy
* Use of central nervous system (CNS) stimulants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (98):
- United States (35):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longmont, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biddeford, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Clair Shores, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southfield, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corvallis, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Georgetown, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakville, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- France (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corbeil-Essonnes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rochelle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mantes-la-Jolie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Narbonne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Mandé
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vénissieux
- Germany (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aschaffenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Lauterberg im Harz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Staffelstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hirschhorn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuwied
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pohlheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotenburg-Fulda
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghaziabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- South Korea (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sungnam-Si
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dos Hermanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiayi City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yung-Kang, Tainan

REFERENCES:
- [Derived] Ferdinand KC, Dunn J, Nicolay C, Sam F, Blue EK, Wang H. Weight-dependent and weight-independent effects of dulaglutide on blood pressure in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):49. doi: 10.1186/s12933-023-01775-x. PMID 36894938
- [Derived] Sherman SI, Kloos RT, Tuttle RM, Pontecorvi A, Volzke H, Harper K, Vance C, Alston JT, Usborne AL, Sloop KW, Lakshmanan M. No calcitonin change in a person taking dulaglutide diagnosed with pre-existing medullary thyroid cancer. Diabet Med. 2018 Mar;35(3):381-385. doi: 10.1111/dme.13437. PMID 28755389
- [Derived] Boustani MA, Pittman I 4th, Yu M, Thieu VT, Varnado OJ, Juneja R. Similar efficacy and safety of once-weekly dulaglutide in patients with type 2 diabetes aged >/=65 and <65 years. Diabetes Obes Metab. 2016 Aug;18(8):820-8. doi: 10.1111/dom.12687. Epub 2016 Jun 7. PMID 27161178
- [Derived] Yu M, Van Brunt K, Varnado OJ, Boye KS. Patient-reported outcome results in patients with type 2 diabetes treated with once-weekly dulaglutide: data from the AWARD phase III clinical trial programme. Diabetes Obes Metab. 2016 Apr;18(4):419-24. doi: 10.1111/dom.12624. Epub 2016 Feb 4. PMID 26691396
- [Derived] Weinstock RS, Guerci B, Umpierrez G, Nauck MA, Skrivanek Z, Milicevic Z. Safety and efficacy of once-weekly dulaglutide versus sitagliptin after 2 years in metformin-treated patients with type 2 diabetes (AWARD-5): a randomized, phase III study. Diabetes Obes Metab. 2015 Sep;17(9):849-58. doi: 10.1111/dom.12479. Epub 2015 May 20. PMID 25912221
- [Derived] Skrivanek Z, Gaydos BL, Chien JY, Geiger MJ, Heathman MA, Berry S, Anderson JH, Forst T, Milicevic Z, Berry D. Dose-finding results in an adaptive, seamless, randomized trial of once-weekly dulaglutide combined with metformin in type 2 diabetes patients (AWARD-5). Diabetes Obes Metab. 2014 Aug;16(8):748-56. doi: 10.1111/dom.12305. Epub 2014 May 22. PMID 24762094
- [Derived] Spencer K, Colvin K, Braunecker B, Brackman M, Ripley J, Hines P, Skrivanek Z, Gaydos B, Geiger MJ. Operational challenges and solutions with implementation of an adaptive seamless phase 2/3 study. J Diabetes Sci Technol. 2012 Nov 1;6(6):1296-304. doi: 10.1177/193229681200600608. PMID 23294774
- See also: (Lilly Clinical Trial Registry) — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- 3.0 mg LY2189265: LY2189265 (Dulaglutide): 3.0 milligrams (mg), subcutaneous (SC) injection, once weekly up to decision point (maximum exposure duration of 24.1 weeks)
  Placebo: tablet, administered orally, once daily up to decision point (maximum exposure duration of 24.1 weeks)
  Metformin: at least 1500 milligrams per day (mg/day), administered orally up to decision point (maximum exposure duration of 24.1 weeks)
- 2.0 mg LY2189265: LY2189265 (Dulaglutide): 2.0 milligrams (mg), subcutaneous (SC) injection, once weekly up to decision point (maximum exposure duration of 20.4 weeks)
  Placebo: tablet, administered orally, once daily up to decision point (maximum exposure duration of 20.4 weeks)
  Metformin: at least 1500 milligrams per day (mg/day), administered orally up to decision point (maximum exposure duration of 20.4 weeks)
- 1.5 mg LY2189265: LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
- 1.0 mg LY2189265: LY2189265 (Dulaglutide): 1.0 milligrams (mg), subcutaneous (SC) injection, once weekly up to decision point (maximum exposure duration of 24.4 weeks)
  Placebo: tablet, administered orally, once daily up to decision point (maximum exposure duration of 24.4 weeks)
  Metformin: at least 1500 milligrams per day (mg/day), administered orally up to decision point (maximum exposure duration of 24.4 weeks)
- 0.75 mg LY2189265: LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
- 0.5 mg LY2189265: LY2189265 (Dulaglutide): 0.5 milligrams (mg), subcutaneous (SC) injection, once weekly up to decision point (maximum exposure duration of 27.4 weeks)
  Placebo: tablet, administered orally, once daily up to decision point (maximum exposure duration of 27.4 weeks)
  Metformin: at least 1500 milligrams per day (mg/day), administered orally up to decision point (maximum exposure duration of 27.4 weeks)
- 0.25 mg LY2189265: LY2189265 (Dulaglutide): 0.25 milligrams (mg), subcutaneous (SC) injection, once weekly up to decision point (maximum exposure duration of 24.4 weeks)
  Placebo: tablet, administered orally, once daily up to decision point (maximum exposure duration of 24.4 weeks)
  Metformin: at least 1500 milligrams per day (mg/day), administered orally up to decision point (maximum exposure duration of 24.4 weeks)
- Placebo/Sitagliptin: Placebo: solution, subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 26 weeks
  Sitagliptin: after 26 weeks, 100-milligrams (mg) tablet, administered orally, once daily for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
Period: Overall Study
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin
Started | 15 | 30 | 304 | 10 | 302 | 25 | 24 | 315 | 177
Received at Least 1 Dose of Study Drug | 15 | 30 | 304 | 10 | 302 | 25 | 24 | 315 | 177
Entered Study Before Dose Decision Point | 15 | 30 | 25 | 10 | 21 | 25 | 24 | 42 | 38
Completed Up to Dose Decision Point | 8 (These participants discontinued the study after the dose decision point.) | 25 (These participants discontinued the study after the dose decision point.) | 24 (These participants continued the study after the dose decision point (selected arm).) | 8 (These participants discontinued the study after the dose decision point.) | 21 (These participants continued the study after the dose decision point (selected arm).) | 21 (These participants discontinued the study after the dose decision point.) | 23 (These participants discontinued the study after the dose decision point.) | 42 (These participants continued the study after the dose decision point (comparator arm).) | 34 (These participants continued the study after the dose decision point (comparator arm).)
Entered Study After Dose Decision Point | 0 | 0 | 279 | 0 | 281 | 0 | 0 | 273 | 139
Completed 26-Week Visit | 0 | 0 | 258 | 2 | 268 | 2 | 2 | 270 | 124
Completed 52-Week Visit | 0 | 0 | 238 | 0 | 243 | 0 | 0 | 238 | 112
Completed | 0 | 0 | 192 | 0 | 184 | 0 | 0 | 186 | 95
Not Completed | 15 | 30 | 112 | 10 | 118 | 25 | 24 | 129 | 82
Not completed — Entry Criteria Not Met | 0 | 0 | 5 | 0 | 3 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 13 | 0 | 11 | 1 | 0 | 9 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 18 | 0 | 24 | 2 | 0 | 36 | 21
Not completed — Physician Decision | 0 | 0 | 4 | 1 | 11 | 0 | 0 | 9 | 9
Not completed — Adverse Event | 4 | 4 | 63 | 1 | 64 | 0 | 1 | 65 | 39
Not completed — Protocol Violation | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 3 | 1
Not completed — Sponsor Decision, Arm Discontinued | 8 | 25 | 0 | 8 | 0 | 21 | 23 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 4 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin | Total
Number analyzed (Participants) | 15 | 30 | 304 | 10 | 302 | 25 | 24 | 315 | 177 | 1202
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.81 (10.66) | 52.56 (10.95) | 53.66 (10.02) | 55.38 (8.71) | 54.35 (9.81) | 54.70 (9.72) | 56.51 (6.56) | 53.75 (10.27) | 54.91 (9.05) | 54.09 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 158 | 7 | 168 | 12 | 15 | 164 | 87 | 643
  Male | 5 | 8 | 146 | 3 | 134 | 13 | 9 | 151 | 90 | 559
Race/Ethnicity, Customized [Number; unit: participants]
  Aboriginal and/or Torres Strait Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  African | 1 | 3 | 16 | 0 | 12 | 2 | 0 | 7 | 9 | 50
  Caucasian | 7 | 13 | 157 | 4 | 162 | 9 | 12 | 158 | 91 | 613
  East Asian | 0 | 6 | 50 | 0 | 47 | 0 | 5 | 52 | 28 | 188
  Hispanic | 7 | 8 | 54 | 6 | 51 | 14 | 6 | 67 | 38 | 251
  Native American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  West Asian (Indian sub-continent) | 0 | 0 | 27 | 0 | 30 | 0 | 1 | 28 | 11 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 17 | 73 | 4 | 83 | 10 | 7 | 80 | 46 | 329
  Taiwan | 0 | 1 | 19 | 0 | 18 | 0 | 3 | 20 | 12 | 73
  Spain | 0 | 0 | 10 | 0 | 11 | 0 | 0 | 11 | 4 | 36
  Russian Federation | 0 | 0 | 21 | 0 | 18 | 0 | 0 | 17 | 8 | 64
  India | 0 | 0 | 27 | 0 | 29 | 0 | 0 | 28 | 12 | 96
  France | 0 | 0 | 12 | 0 | 14 | 0 | 0 | 12 | 8 | 46
  Mexico | 3 | 3 | 32 | 5 | 30 | 10 | 6 | 35 | 27 | 151
  Puerto Rico | 1 | 2 | 12 | 0 | 5 | 3 | 0 | 10 | 7 | 40
  Canada | 0 | 0 | 13 | 0 | 11 | 0 | 0 | 12 | 6 | 42
  Poland | 1 | 0 | 20 | 0 | 23 | 2 | 2 | 23 | 12 | 83
  Romania | 1 | 2 | 7 | 1 | 4 | 0 | 4 | 8 | 5 | 32
  Germany | 0 | 0 | 31 | 0 | 31 | 0 | 0 | 28 | 15 | 105
  Korea, Republic of | 0 | 5 | 27 | 0 | 25 | 0 | 2 | 31 | 15 | 105
Body Weight [Mean (Standard Deviation); unit: kilograms] | 85.09 (14.25) | 86.56 (18.33) | 86.67 (17.45) | 89.48 (18.06) | 86.22 (17.99) | 88.84 (14.98) | 81.94 (17.67) | 85.97 (16.91) | 87.07 (16.86) | 86.38 (17.28)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 31.02 (4.69) | 31.45 (4.88) | 31.40 (4.57) | 33.89 (4.44) | 31.15 (4.44) | 32.53 (4.61) | 31.06 (3.94) | 31.02 (4.20) | 31.37 (4.25) | 31.27 (4.39)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7.95 (1.11) | 8.36 (1.04) | 8.12 (1.05) | 7.87 (0.62) | 8.19 (1.11) | 8.30 (1.34) | 7.82 (0.80) | 8.09 (1.09) | 8.10 (1.14) | 8.13 (1.09)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.79 (6.34) | 6.92 (5.12) | 6.95 (5.50) | 7.04 (4.57) | 7.34 (4.92) | 6.75 (3.99) | 6.74 (4.20) | 7.16 (4.89) | 6.96 (5.43) | 7.09 (5.12)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: millimoles per liter (mmol/L)] | NA (NA) — Baseline fasting plasma glucose was not summarized for this treatment arm. | NA (NA) — Baseline fasting plasma glucose was not summarized for this treatment arm. | 9.75 (3.27) | NA (NA) — Baseline fasting plasma glucose was not summarized for this treatment arm. | 9.68 (2.94) | NA (NA) — Baseline fasting plasma glucose was not summarized for this treatment arm. | NA (NA) — Baseline fasting plasma glucose was not summarized for this treatment arm. | 9.56 (2.80) | 9.86 (3.15) | NA (NA) — Total Mean (SD) were not calculated for this baseline measure.

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin (HbA1c) Change From Baseline
Description: Least squares (LS) means were calculated using analysis of covariance (ANCOVA) and last observation carried forward (LOCF) imputation with country and treatment as fixed effects and baseline HbA1c as a covariate.
Time Frame: Baseline, 52 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and active comparator (Sitagliptin) arms who had evaluable HbA1c data. Last observation carried forward was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 301 | 297 | 311
percentage of HbA1c | -1.10 (0.06) | -0.87 (0.06) | -0.39 (0.06)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Power was estimated at approximately 89% based on a simulation study using the "most likely" pharmacodynamic model, assuming a 20% drop out rate (missing completely at random) at 52 weeks and enrollment of 5 participants per week. A predictive power calculation was planned to select either 263 or 333 as the minimum total sample size needed (sum of Stage 1 and 2) per arm. If the predictive power of the higher LY2189265 dose based on 263 participants in total exceeded 85%, then 263 would be used; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying gatekeeping strategies; p < 0.001, ANCOVA — P-value is adjusted for multiplicity, based on tree-gatekeeping strategy. To determine significance, p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.71, 95% CI 2-sided [-0.87 to -0.55]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Sitagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying a gatekeeping strategy; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.63 to -0.31]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.71, 95% CI 2-sided [-0.87 to -0.55]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.63 to -0.31]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at the Dose Decision Point
Description: Change from baseline in HbA1c was 1 of the 4 measures included in the clinical utility index (CUI) used to evaluate the dose decision. The maximum duration of exposure to LY2189265, Sitagliptin, or Placebo (across all treatment arms) at the decision point was 27.4 weeks.
Time Frame: Baseline up to 27.4 weeks
Population: All participants randomized before the dose decision point who had evaluable HbA1c data.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Placebo/Sitagliptin (Baseline Through 26 Weeks): Placebo: solution, subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 26 weeks
  Sitagliptin: after 26 weeks, 100-milligrams (mg) tablet, administered orally, once daily for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 10 | 26 | 20 | 8 | 20 | 21 | 14 | 30 | 28
percentage of HbA1c | -1.09 (0.77) | -1.25 (0.68) | -1.49 (1.12) | -0.98 (0.47) | -1.02 (0.99) | -0.94 (0.65) | -0.70 (0.49) | -0.76 (0.86) | -0.06 (0.64)

3. Secondary Outcome: Glycosylated Hemoglobin (HbA1c) Change From Baseline
Description: as for outcome 1
Time Frame: Baseline, 26 weeks, 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable HbA1c data. Last observation carried forward was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 301 | 297 | 311 | 176
percentage of HbA1c
  26 Weeks | -1.22 (0.05) | -1.01 (0.06) | -0.61 (0.05) | 0.03 (0.07)
  104 Weeks | -0.99 (0.06) | -0.71 (0.07) | -0.32 (0.06) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 26 weeks. P-value adjusted for multiplicity based on tree-gatekeeping strategy. To determine significance, p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -1.26, 95% CI 2-sided [-1.42 to -1.09]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = -1.05, 95% CI 2-sided [-1.21 to -0.88]
Statistical Analysis 3: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 26 weeks. One-sided raw p-value with no adjustment for multiplicity; LS Mean Difference = -0.64, 95% CI 2-sided [-0.81 to -0.48]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate was controlled by applying a gatekeeping strategy; p < 0.001, ANCOVA — Comparison at 104 weeks. P-value adjusted for multiplicity based on tree-gatekeeping strategy. To determine significance, p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.67, 95% CI 2-sided [-0.84 to -0.50]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Non-Inferiority or Equivalence — Family-wise Type I error rate controlled by applying gatekeeping strategy; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 4]; LS Mean Difference = -0.39, 95% CI 2-sided [-0.56 to -0.22]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 4]; LS Mean Difference = -0.67, 95% CI 2-sided [-0.84 to -0.50]
Statistical Analysis 7: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 4]; LS Mean Difference = -0.39, 95% CI 2-sided [-0.56 to -0.22]

4. Secondary Outcome: Durability of Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Durability of effect on HbA1c was assessed by comparing the differences in mean change from baseline in HbA1c at 1 time point versus an earlier time point. Least squares (LS) means of change from baseline HbA1c data were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 13, 26, 52, and 104 weeks
Population: All participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms randomized after the dose decision point who had evaluable HbA1c data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 303 | 302 | 314 | 177
percentage of HbA1c
  26 Weeks Versus 13 Weeks (n=269, 269, 276, 136) | -0.03 (0.04) | 0.02 (0.04) | 0.00 (0.04) | -0.14 (0.05)
  52 Weeks Versus 26 Weeks (n=245, 254, 250) | 0.14 (0.05) | 0.16 (0.05) | 0.24 (0.05) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  104 Weeks Versus 52 Weeks (n=194, 191, 190) | 0.13 (0.06) | 0.16 (0.06) | 0.09 (0.06) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.

5. Secondary Outcome: Fasting Blood Glucose Change From Baseline
Description: Least squares (LS) means of change from baseline were calculated using mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable fasting plasma glucose data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 297 | 296 | 308 | 176
millimoles per liter (mmol/L)
  26 Weeks (n=265, 271, 276, 135) | -2.38 (0.12) | -1.97 (0.12) | -0.97 (0.11) | -0.49 (0.16)
  52 Weeks (n=239, 247, 244) | -2.38 (0.13) | -1.63 (0.13) | -0.90 (0.13) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  104 Weeks (n=190, 187, 181) | -1.99 (0.15) | -1.39 (0.15) | -0.47 (0.15) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Comparison at 26 weeks; LS Mean Difference = -1.89, 95% CI 2-sided [-2.27 to -1.51]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = -1.48, 95% CI 2-sided [-1.85 to -1.10]
Statistical Analysis 3: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = -0.48, 95% CI 2-sided [-0.86 to -0.11]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 52 weeks; LS Mean Difference = -1.47, 95% CI 2-sided [-1.82 to -1.13]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 52 weeks; LS Mean Difference = -0.73, 95% CI 2-sided [-1.07 to -0.39]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 104 weeks; LS Mean Difference = -1.51, 95% CI 2-sided [-1.93 to -1.10]
Statistical Analysis 7: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 104 weeks; LS Mean Difference = -0.92, 95% CI 2-sided [-1.33 to -0.51]

6. Secondary Outcome: Fasting Insulin Change From Baseline
Description: Least squares (LS) means of change from baseline fasting insulin data were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 104 weeks
Population: All participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms randomized after the dose decision point who had evaluable fasting insulin data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: picomoles per liter (pmol/L)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 254 | 261 | 247 | 122
picomoles per liter (pmol/L)
  26 Weeks (n=238, 249, 230, 115) | 11.59 (6.57) | 10.15 (6.51) | 8.48 (6.68) | -6.92 (9.24)
  52 Weeks (n=207, 218, 200) | 10.57 (5.95) | 12.95 (5.88) | 4.18 (6.01) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  104 Weeks (n=187, 200, 183) | 11.36 (7.58) | 21.56 (7.40) | 0.29 (7.64) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.095, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = 18.51, 95% CI 2-sided [-3.25 to 40.28]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.121, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = 17.08, 95% CI 2-sided [-4.54 to 38.69]
Statistical Analysis 3: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.167, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = 15.41, 95% CI 2-sided [-6.47 to 37.29]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.430, Mixed Models Analysis — Comparison at 52 weeks; LS Mean Difference = 6.38, 95% CI 2-sided [-9.49 to 22.26]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.273, Mixed Models Analysis — Comparison at 52 weeks; LS Mean Difference = 8.77, 95% CI 2-sided [-6.94 to 24.47]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.291, Mixed Models Analysis — Comparison at 104 weeks; LS Mean Difference = 11.07, 95% CI 2-sided [-9.49 to 31.64]
Statistical Analysis 7: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — Comparison at 104 weeks; LS Mean Difference = 21.28, 95% CI 2-sided [1.03 to 41.53]

7. Secondary Outcome: Change From Baseline in Body Weight at Dose Decision Point
Description: Change from baseline in body weight was 1 of the 4 measures included in the clinical utility index (CUI) used to evaluate the dose decision. The maximum duration of exposure to LY2189265, Sitagliptin, or Placebo (across all treatment arms) at the decision point was 27.4 weeks.
Time Frame: Baseline up to 27.4 weeks
Population: All participants randomized before the dose decision point who had evaluable body weight data.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 14 | 30 | 23 | 9 | 20 | 22 | 17 | 35 | 33
kilograms (kg) | -3.32 (3.37) | -2.15 (1.97) | -2.12 (1.93) | -2.23 (1.63) | -1.17 (2.30) | -1.53 (1.88) | -0.85 (1.47) | -0.43 (1.78) | -0.56 (1.69)

8. Secondary Outcome: Body Weight Change From Baseline
Description: Least squares (LS) means of change from baseline body weight were calculated using analysis of covariance (ANCOVA) and last observation carried forward (LOCF) imputation with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable body weight data. Last observation carried forward was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 303 | 299 | 314 | 177
kilograms (kg)
  26 Weeks | -3.18 (0.18) | -2.63 (0.19) | -1.46 (0.18) | -1.47 (0.24)
  52 Weeks | -3.03 (0.22) | -2.60 (0.23) | -1.53 (0.22) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  104 Weeks | -2.88 (0.25) | -2.39 (0.26) | -1.75 (0.25) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 26 weeks; LS Mean Difference = -1.70, 95% CI 2-sided [-2.27 to -1.14]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 26 weeks; LS Mean Difference = -1.16, 95% CI 2-sided [-1.73 to -0.60]
Statistical Analysis 3: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.953, ANCOVA — Comparison at 26 weeks; LS Mean Difference = 0.02, 95% CI 2-sided [-0.54 to 0.58]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 52 weeks; LS Mean Difference = -1.50, 95% CI 2-sided [-2.08 to -0.92]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 52 weeks; LS Mean Difference = -1.07, 95% CI 2-sided [-1.65 to -0.48]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, ANCOVA — Comparison at 104 weeks; LS Mean Difference = -1.14, 95% CI 2-sided [-1.78 to -0.49]
Statistical Analysis 7: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.054, ANCOVA — Comparison at 104 weeks; LS Mean Difference = -0.64, 95% CI 2-sided [-1.29 to 0.01]

9. Secondary Outcome: Durability of Change From Baseline Body Weight
Description: Durability of effect on body weight was assessed by comparing the differences in mean change from baseline in body weight at 1 time point versus an earlier time point. Least squares (LS) means of change from baseline body weight data were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 13, 26, 52, and 104 weeks
Population: All participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms randomized after the dose decision point who had evaluable body weight data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
kilograms (kg)
  26 Weeks Versus 13 Weeks (n=271, 278, 282, 138) | -0.53 (0.14) | -0.57 (0.14) | -0.42 (0.13) | -0.37 (0.18)
  52 Weeks Versus 26 Weeks (n=246, 255, 253) | 0.17 (0.18) | 0.06 (0.18) | -0.04 (0.18) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  104 Weeks Versus 26 Weeks (n=197, 192, 191) | 0.42 (0.23) | 0.32 (0.24) | -0.39 (0.23) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.

10. Secondary Outcome: Waist Circumference Change From Baseline
Description: Least squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable waist circumference data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 299 | 301 | 312 | 175
centimeters (cm)
  26 Weeks (n=266, 273, 277, 138) | -2.89 (0.24) | -1.78 (0.24) | -1.45 (0.24) | -1.20 (0.32)
  52 Weeks (n=238, 250, 247) | -2.91 (0.29) | -2.05 (0.29) | -1.45 (0.29) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  104 Weeks (n=192, 189, 188) | -2.57 (0.35) | -1.75 (0.35) | -1.20 (0.35) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = -1.69, 95% CI 2-sided [-2.45 to -0.93]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.133, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = -0.58, 95% CI 2-sided [-1.34 to 0.18]
Statistical Analysis 3: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.512, Mixed Models Analysis — Comparison at 26 weeks; LS Mean Difference = -0.25, 95% CI 2-sided [-1.01 to 0.50]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Comparison at 52 weeks; LS Mean Difference = -1.46, 95% CI 2-sided [-2.23 to -0.69]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis — Comparison at 52 weeks; LS Mean Difference = -0.59, 95% CI 2-sided [-1.36 to 0.17]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — Comparison at 104 weeks; LS Mean Difference = -1.36, 95% CI 2-sided [-2.30 to -0.42]
Statistical Analysis 7: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p = 0.256, Mixed Models Analysis — Comparison at 104 weeks; LS Mean Difference = -0.54, 95% CI 2-sided [-1.48 to 0.40]

11. Secondary Outcome: Percentage of Participants Who Achieve Glycosylated Hemoglobin (HbA1c) <7% or ≤6.5%
Description: The percentage of participants achieving HbA1c levels <7.0% and ≤6.5% was analyzed using a logistic regression model and last observation carried forward (LOCF) imputation with baseline, country, and treatment as factors included in the model.
Time Frame: Baseline, 26, 52, and 104 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 302 | 297 | 312 | 176
percentage of participants
  <7.0% at 26 Weeks | 60.9 | 55.2 | 37.8 | 21.0
  <7.0% at 52 Weeks | 57.6 | 48.8 | 33.0 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  <7.0% at 104 Weeks | 54.3 | 44.8 | 31.1 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  ≤6.5% at 26 Weeks | 46.7 | 31.0 | 21.8 | 12.5
  ≤6.5% at 52 Weeks | 41.7 | 29.0 | 19.2 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  ≤6.5% at 104 Weeks | 39.1 | 24.2 | 14.1 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 26 weeks; Odds Ratio (OR) = 11.3, 95% CI 2-sided [6.8 to 18.8]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 26 weeks; Odds Ratio (OR) = 8.6, 95% CI 2-sided [5.2 to 14.3]
Statistical Analysis 3: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 26 weeks; Odds Ratio (OR) = 3.0, 95% CI 2-sided [1.8 to 4.8]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 52 weeks; Odds Ratio (OR) = 4.0, 95% CI 2-sided [2.7 to 5.9]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 52 weeks; Odds Ratio (OR) = 2.7, 95% CI 2-sided [1.8 to 3.9]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 104 weeks; Odds Ratio (OR) = 3.4, 95% CI 2-sided [2.4 to 5.0]
Statistical Analysis 7: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c <7.0% at 104 weeks; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.6 to 3.3]
Statistical Analysis 8: Comparison: 1.5 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c ≤6.5% at 26 weeks; Odds Ratio (OR) = 11.5, 95% CI 2-sided [6.5 to 20.4]
Statistical Analysis 9: Comparison: 0.75 mg LY2189265 vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c ≤6.5% at 26 weeks; Odds Ratio (OR) = 5.0, 95% CI 2-sided [2.8 to 8.8]
Statistical Analysis 10: Comparison: Sitagliptin vs Placebo/Sitagliptin (Baseline Through 26 Weeks); Test type: Superiority or Other; p = 0.005, Regression, Logistic — Comparison of HbA1c ≤6.5 at 26 weeks; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.3 to 4.1]
Statistical Analysis 11: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c ≤6.5% at 52 weeks; Odds Ratio (OR) = 4.4, 95% CI 2-sided [2.9 to 6.8]
Statistical Analysis 12: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c ≤6.5% at 52 weeks; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.5 to 3.5]
Statistical Analysis 13: Comparison: 1.5 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c ≤6.5% at 104 weeks; Odds Ratio (OR) = 5.2, 95% CI 2-sided [3.4 to 7.9]
Statistical Analysis 14: Comparison: 0.75 mg LY2189265 vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Comparison of HbA1c ≤6.5% at 104 weeks; Odds Ratio (OR) = 2.4, 95% CI 2-sided [1.5 to 3.7]

12. Secondary Outcome: Incidence of Hypoglycemic Episodes
Description: Hypoglycemic episodes (HE) were classified as severe (defined as episodes requiring assistance from another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia and has a plasma glucose level of ≤3.9 millimoles per liter [mmol/L]), asymptomatic (defined as episodes not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of ≤3.9 mmol/L), nocturnal (defined as any episode that occurred between bedtime and waking), or probable symptomatic (defined as episodes during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The number of participants with self-reported hypoglycemic events is summarized cumulatively.
Time Frame: Baseline through 26 and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
participants
  Severe HE, 26 Weeks | 0 | 0 | 0 | 0
  Severe HE, 104 Weeks | 0 | 0 | 0 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Documented Symptomatic HE, 26 Weeks | 17 | 8 | 10 | 2
  Documented Symptomatic HE, 104 Weeks | 33 | 19 | 18 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Asymptomatic HE, 26 Weeks | 5 | 5 | 0 | 0
  Asymptomatic HE, 104 Weeks | 9 | 9 | 3 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Nocturnal HE, 26 Weeks | 7 | 5 | 2 | 0
  Nocturnal HE, 104 Weeks | 14 | 13 | 10 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Probable HE, 26 Weeks | 5 | 0 | 2 | 0
  Probable HE, 104 Weeks | 6 | 2 | 6 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.

13. Secondary Outcome: Rate of Hypoglycemic Episodes
Description: Hypoglycemic episodes (HE) were classified as severe (defined as episodes requiring assistance from another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia and has a plasma glucose level of ≤3.9 millimoles per liter [mmol/L]), asymptomatic (defined as episodes not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of ≤3.9 mmol/L), nocturnal (defined as any episode that occurred between bedtime and waking), or probable symptomatic (defined as episodes during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The 1-year adjusted rate of HE is summarized cumulatively.
Time Frame: Baseline through 26 and 104 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
episodes per participant per year
  Severe HE, 26 Weeks | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Severe HE, 104 Weeks | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Documented Symptomatic HE, 26 Weeks | 0.3 (1.5) | 0.1 (0.9) | 0.1 (0.7) | 0.1 (0.9)
  Documented Symptomatic HE, 104 Weeks | 0.2 (0.9) | 0.2 (1.9) | 0.2 (1.4) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Asymptomatic HE, 26 Weeks | 0.1 (0.8) | 0.1 (0.5) | 0.0 (0.0) | 0.0 (0.0)
  Asymptomatic HE, 104 Weeks | 0.1 (0.4) | 0.0 (0.2) | 0.0 (0.1) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Nocturnal HE, 26 Weeks | 0.1 (0.9) | 0.1 (0.6) | 0.0 (0.4) | 0.0 (0.0)
  Nocturnal HE, 104 Weeks | 0.1 (0.5) | 0.0 (0.2) | 0.1 (0.5) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Probable Symptomatic HE, 26 Weeks | 0.0 (0.4) | 0.0 (0.0) | 0.0 (0.2) | 0.0 (0.0)
  Probable Symptomatic HE, 104 Weeks | 0.0 (0.1) | 0.0 (0.0) | 0.0 (0.1) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.

14. Secondary Outcome: Beta Cell Function and Insulin Sensitivity (HOMA2)
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta (β)-cell function. HOMA2-%B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state beta cell function (%B) as a percentage of a normal reference population (normal young adults). HOMA2-%S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S), as percentages of a normal reference population (normal young adults). The normal reference population for both HOMA2-%B and HOMA2-%S were set at 100%. Least squares (LS) means of change from baseline of C-peptide based HOMA2-%B and HOMA2-%S were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26, 52, and 104 weeks
Population: All participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms randomized after the dose decision point and who had evaluable HOMA2 data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: HOMA2-%
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 242 | 251 | 238 | 115
HOMA2-%
  HOMA2-%B, 26 Weeks (n=206, 226, 206, 84) | 32.28 (2.67) | 26.98 (2.60) | 10.81 (2.66) | 1.60 (4.02)
  HOMA2-%B, 52 Weeks (n=188, 198, 180) | 33.57 (2.51) | 22.30 (2.47) | 6.66 (2.53) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  HOMA2-%B, 104 Weeks (n=148, 154, 134) | 30.89 (3.05) | 19.11 (3.00) | 1.47 (3.15) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  HOMA2-%S, 26 Weeks (n=206, 226, 206, 84) | 5.75 (2.34) | 0.78 (2.28) | 2.29 (2.33) | 9.82 (3.50)
  HOMA2-%S, 52 Weeks (n=188, 198, 180) | 4.69 (2.35) | 2.28 (2.32) | 4.25 (2.37) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.
  HOMA2-%S, 104 Weeks (n=148, 154, 134) | 3.82 (3.00) | -0.12 (2.95) | 5.61 (3.11) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for participants who received Placebo at this time point.

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events at 26 Weeks
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with 1 or more TEAEs is summarized cumulatively. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
participants | 208 | 204 | 185 | 111

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events at 52 Weeks
Description: as for outcome 15
Time Frame: Baseline through 52 weeks
Population: All randomized participants in the LY2189265 and active comparator (Sitagliptin) arms.
Measure: Number; unit: participants
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 15 | 30 | 304 | 10 | 302 | 25 | 24 | 315
participants | 9 | 20 | 233 | 8 | 231 | 15 | 10 | 219

17. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events at 104 Weeks
Description: as for outcome 15
Time Frame: Baseline through 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and active comparator (Sitagliptin) arms.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 304 | 302 | 315
participants | 259 | 255 | 242

18. Secondary Outcome: Number of Participants With Treatment-emergent Abnormal Laboratory Tests at 26 Weeks
Description: The number of participants with treatment-emergent abnormal laboratory results (defined as abnormalities that first occur after baseline) was summarized cumulatively for alkaline phosphatase, alanine aminotransferase or serum glutamic pyruvic transaminase (ALT/SGPT), amylase (pancreatic and total), aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST/SGOT), basophils, bilirubin (direct and total), calcitonin, chloride, creatine phosphokinase (CPK), creatinine, creatinine clearance, eosinophils, erythrocytes, gamma glutamyltransferase (GGT), hematocrit, hemoglobin, leukocytes, lipase, lymphocytes, mean cell hemoglobin concentration (MCHC), mean cell volume (MCV), monocytes, neutrophils, platelets, potassium, sodium, urea nitrogen, and urine microalbumin-to-creatinine ratio (UMCR).
Time Frame: Baseline through 26 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms with baseline value not in the specified direction of treatment-emergent abnormality and at least 1 postbaseline result.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
participants
  Alkaline Phosphatase (n=276, 258, 281, 162) | 9 | 3 | 12 | 3
  ALT/SGPT (n=232, 237, 244, 128) | 18 | 24 | 25 | 8
  Amylase Pancreatic, High (n=283, 277, 295, 160) | 54 | 55 | 42 | 18
  Amylase Total (n=266, 265, 277, 143) | 33 | 33 | 27 | 13
  AST/SGOT (n=273, 269, 284, 148) | 14 | 12 | 18 | 7
  Basophils, High (n=268, 259, 278, 163) | 1 | 0 | 1 | 0
  Basophils, Low (n=269, 259, 278, 163) | 0 | 0 | 0 | 0
  Bilirubin Direct, High (n=295, 291, 307, 171) | 1 | 1 | 1 | 2
  Bilirubin Total, High (n=295, 290, 305, 168) | 2 | 4 | 4 | 1
  Calcitonin, High (n=226, 233, 230, 113) | 1 | 2 | 2 | 0
  Chloride, High (n=299, 293, 310, 174) | 0 | 1 | 0 | 0
  Chloride, Low (n=299, 293, 308, 174) | 1 | 2 | 1 | 1
  CPK, High (n=273, 262, 276, 156 | 29 | 20 | 30 | 7
  Creatinine, High (n=294, 285, 303, 172) | 7 | 10 | 5 | 5
  Creatinine Clearance, High (n=164, 186, 180, 107) | 17 | 28 | 26 | 25
  Creatinine Clearance, Low (n=292, 278,303,168) | 11 | 17 | 12 | 6
  Eosinophils, High (n=258, 256, 275, 157) | 4 | 11 | 6 | 2
  Eosinophils, Low (n=269, 259, 278, 163) | 0 | 0 | 0 | 0
  Erythrocyte Count, High (n=279, 272, 287, 164) | 1 | 1 | 0 | 0
  Erythrocyte Count, Low (n=274, 268, 280, 161) | 12 | 7 | 7 | 3
  GGT, High (n=234, 240, 245, 144) | 9 | 11 | 23 | 10
  Hematocrit, High (n=273, 265, 279, 161) | 1 | 1 | 1 | 2
  Hematocrit, Low (n=256, 242, 259, 157) | 13 | 10 | 6 | 5
  Hemoglobin, High (n=278, 271, 289, 164) | 1 | 1 | 1 | 2
  Hemoglobin, Low (n=262, 249, 265, 162) | 13 | 16 | 5 | 3
  Leukocyte Count, High (n=272, 265, 286, 165) | 3 | 6 | 1 | 0
  Leukocyte Count, Low (n=272, 262, 280, 165) | 2 | 3 | 4 | 1
  Lipase, High (n=255, 248, 269, 147) | 109 | 92 | 97 | 37
  Lymphocytes, High (n=249, 253, 269, 161) | 5 | 9 | 6 | 3
  Lymphocytes, Low (n=265, 258, 273, 159) | 3 | 3 | 4 | 2
  MCHC, High (n=274, 265, 280, 163) | 0 | 0 | 0 | 0
  MCHC, Low (n=273, 263, 279, 163) | 0 | 2 | 0 | 0
  MCV, High (n=261, 248, 263, 156) | 19 | 12 | 14 | 5
  MCV, Low (n=264, 252, 275, 162) | 3 | 2 | 2 | 0
  Monocytes, High (n=266, 258, 274, 163) | 1 | 0 | 3 | 1
  Monocytes, Low (n=265, 255, 274, 158) | 6 | 5 | 8 | 10
  Neutrophils, High (n=264, 255, 276, 161) | 4 | 5 | 3 | 1
  Neutrophils, Low (n=263, 251, 271, 162) | 2 | 1 | 2 | 1
  Platelet Count, High (n=265, 260, 281, 160) | 0 | 0 | 1 | 0
  Platelet Count, Low (n=262, 252, 269, 154) | 2 | 3 | 6 | 3
  Potassium, High (n=297, 291, 307, 172) | 7 | 2 | 5 | 4
  Potassium, Low (n=298, 293, 308, 169) | 4 | 6 | 3 | 1
  Sodium, High (n=291, 291, 307, 170) | 3 | 4 | 4 | 4
  Sodium, Low (n=298, 292, 305, 174) | 2 | 1 | 4 | 1
  Urea Nitrogen, High (n=287, 282, 305, 169) | 11 | 17 | 13 | 5
  UMCR, High (n=217, 204, 232, 130) | 18 | 9 | 13 | 5

19. Secondary Outcome: Number of Participants With Treatment-emergent Abnormal Laboratory Tests at 52 Weeks
Description: The number of participants with treatment-emergent abnormal laboratory results (defined as abnormalities that first occur after baseline) was summarized cumulatively for alkaline phosphatase, alanine aminotransferase or serum glutamic pyruvic transaminase (ALT/SGPT), amylase (pancreatic and total), aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST/SGOT), basophils, bilirubin (direct and total), calcitonin, chloride, creatine phosphokinase (CPK), creatinine, creatinine clearance, eosinophils, erythrocytes, gamma glutamyltransferase (GGT), hematocrit, hemoglobin, leukocytes, lipase, lymphocytes, mean cell hemoglobin concentration (MCHC), mean cell volume (MCV), monocytes, neutrophils, platelets, potassium, sodium, urea nitrogen, and urine microalbumin-to-creatinine ratio (UMCR) .
Time Frame: Baseline through 52 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and active comparator (Sitagliptin) arms with baseline value not in the specified direction of treatment-emergent abnormality and at least 1 postbaseline result.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 304 | 302 | 315
participants
  Alkaline Phosphatase, High (n=276, 258, 281) | 10 | 6 | 16
  ALT/SGPT, High (n=232, 237, 244) | 25 | 27 | 28
  Amylase Pancreatic, High (n=283, 277, 295) | 67 | 70 | 55
  Amylase Total, High (n=266, 265, 277) | 38 | 42 | 36
  AST/SGOT, High (n=273, 269, 284) | 15 | 19 | 25
  Basophils, High (n=276, 268, 287) | 1 | 0 | 1
  Basophils, Low (n=277, 268, 287) | 0 | 0 | 0
  Bilirubin Direct, High (n=295, 291, 307) | 1 | 1 | 2
  Bilirubin Total, High (n=295, 290, 305) | 2 | 6 | 5
  Calcitonin, High (n=233, 239, 235) | 4 | 2 | 2
  Chloride, High (n=299, 293, 310) | 0 | 1 | 0
  Chloride, Low (n=299, 293, 308) | 1 | 2 | 2
  CPK, High (n=273, 262, 276) | 38 | 28 | 43
  Creatinine, High (n=294, 285, 303) | 9 | 10 | 6
  Creatinine Clearance, High (n=164, 186, 180) | 23 | 30 | 29
  Creatinine Clearance, Low (n=292, 278, 303) | 18 | 20 | 15
  Eosinophils, High (n=265, 265, 283) | 11 | 14 | 10
  Eosinophils, Low (n=277, 268, 287) | 0 | 0 | 0
  Erythrocyte Count, High (n=283, 276, 292) | 3 | 1 | 1
  Erythrocyte Count, Low (n=278, 272, 285) | 15 | 9 | 11
  GGT, High (n=234, 240, 245) | 10 | 14 | 34
  Hematocrit, High (n=280, 274, 290) | 3 | 2 | 2
  Hematocrit, Low (n=262, 251, 269) | 21 | 13 | 11
  Hemoglobin, High (n=282, 275, 294) | 3 | 1 | 1
  Hemoglobin, Low (n=265, 253, 269) | 21 | 19 | 11
  Leukocyte Count, High (n=277, 270, 292) | 7 | 6 | 3
  Leukocyte Count, Low (n=277, 267, 284) | 5 | 3 | 9
  Lipase, High (n=255, 248, 269) | 124 | 111 | 110
  Lymphocytes, High (n=257, 262, 278) | 12 | 15 | 11
  Lymphocytes, Low (n=273, 266, 280) | 4 | 4 | 11
  MCHC, High (n=281, 274, 291) | 0 | 0 | 0
  MCHC, Low (n=280, 272, 290) | 2 | 3 | 3
  MCV, High (n=267, 256, 273) | 25 | 18 | 19
  MCV, Low (n=270, 261, 286) | 3 | 2 | 4
  Monocytes, High (n=274, 267, 283) | 1 | 0 | 5
  Monocytes, Low (n=271, 264, 282) | 8 | 9 | 15
  Neutrophils, High (n=272, 263, 285) | 8 | 7 | 7
  Neutrophils, Low (n=271, 260, 279) | 6 | 2 | 6
  Platelet Count, High (n=272, 267, 287) | 0 | 2 | 2
  Platelet Count, Low (n=269, 259, 275) | 4 | 5 | 8
  Potassium, High (n=297, 291, 307) | 10 | 5 | 5
  Potassium, Low (n=298, 293, 308) | 6 | 7 | 5
  Sodium, High (n=291, 291, 307) | 5 | 8 | 4
  Sodium, Low (n=298, 292, 305) | 3 | 1 | 4
  Urea Nitrogen, High (n=287, 282, 305) | 14 | 19 | 21
  UMCR, High (n=223, 212, 238) | 33 | 21 | 18

20. Secondary Outcome: Number of Participants With Treatment-emergent Abnormal Laboratory Tests at 104 Weeks
Description: as for outcome 18
Time Frame: Baseline through 104 weeks
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 304 | 302 | 315
participants
  Alkaline Phosphate, High (n=276, 258, 281) | 13 | 11 | 20
  ALT/SGPT, High (n=232, 237, 244) | 29 | 37 | 39
  Amylase Pancreatic, High (n=283, 277, 295) | 81 | 78 | 61
  Amylase Total, High (n=266, 265, 277) | 44 | 55 | 43
  AST/SGOT, High (n=273, 269, 284) | 21 | 27 | 36
  Basophils, High (n=276, 268, 288) | 1 | 0 | 1
  Basophils, Low (n=277, 268, 288) | 0 | 0 | 0
  Bilirubin Direct, High (n=295, 291, 307) | 2 | 1 | 3
  Bilirubin Total, High (n=295, 290, 305) | 3 | 8 | 6
  Calcitonin, High (n=233, 239, 235) | 5 | 3 | 4
  Chloride, High (n=299, 293, 310) | 0 | 2 | 1
  Chloride, Low (n=299, 293, 308) | 3 | 2 | 3
  CPK, High (n=273, 262, 276) | 52 | 41 | 54
  Creatinine, High (n=294, 285, 303) | 11 | 16 | 9
  Creatinine Clearance, High (n=164, 186, 180) | 26 | 32 | 34
  Creatinine Clearance, Low (n=292, 278, 303) | 24 | 25 | 20
  Eosinophils, High (n=265, 265, 284) | 12 | 22 | 14
  Eosinophils, Low (n=277, 268, 288) | 0 | 0 | 0
  Erythrocyte Count, High (n=283, 276, 292) | 3 | 2 | 1
  Erythrocyte Count, Low (n=278, 272, 285) | 18 | 14 | 19
  GGT, High (n=234, 240, 245) | 16 | 24 | 45
  Hematocrit, High (n=280, 274, 290) | 3 | 6 | 3
  Hematocrit, Low (n=262, 251, 269) | 30 | 24 | 29
  Hemoglobin, High (n=282, 275, 294) | 4 | 3 | 2
  Hemoglobin, Low (n=265, 253, 269) | 30 | 28 | 25
  Leukocyte Count, High (n=277, 270, 292) | 13 | 9 | 8
  Leukocyte Count, Low (n=277, 267, 284) | 9 | 7 | 14
  Lipase, High (n=255, 248, 269) | 142 | 132 | 126
  Lymphocytes, High (n=257, 262, 279) | 19 | 20 | 21
  Lymphocytes, Low (n=273, 266, 281) | 5 | 9 | 12
  MCHC, High (n=281, 274, 291) | 0 | 0 | 0
  MCHC, Low (n=280, 272, 290) | 5 | 4 | 5
  MCV, High (n=267, 256, 273) | 39 | 25 | 25
  MCV, Low (n=270, 261, 286) | 9 | 3 | 4
  Monocytes, High (n=274, 267, 284) | 3 | 1 | 11
  Monocytes, Low (n=271, 264, 283) | 10 | 14 | 17
  Neutrophils, High (n=272, 263, 286) | 15 | 12 | 13
  Neutrophils, Low (n=271, 260, 280) | 10 | 6 | 10
  Platelet Count, High (n=273, 268, 287) | 2 | 3 | 3
  Platelet Count, Low (n=270, 260, 275) | 8 | 7 | 8
  Potassium, High (n=297, 291, 307) | 14 | 9 | 8
  Potassium, Low (n=298, 293, 308) | 8 | 8 | 5
  Sodium, High (n=291, 291, 307) | 10 | 10 | 6
  Sodium, Low (n=298, 292, 305) | 5 | 1 | 5
  Urea Nitrogen, High (n=287, 282, 305) | 17 | 29 | 29
  UMCR, High (n=223, 212, 239) | 38 | 27 | 30

21. Secondary Outcome: Number of Participants With Treatment-emergent Abnormal Lipid Tests
Description: The number of participants with treatment-emergent abnormal lipid test (cholesterol, high density lipoprotein cholesterol [HDL-C], low density lipoprotein cholesterol [LDL-C], and triglycerides [TG]) results (defined as lipid test abnormalities that first occurred after baseline) is summarized cumulatively.
Time Frame: Baseline through 26 and 104 weeks
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
participants
  Cholesterol, High, 26 Weeks (n=144, 158, 139, 58) | 16 | 21 | 20 | 8
  Cholesterol, High, 104 Weeks (n=151, 164, 146) | 34 | 29 | 34 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  HDL-C, High, 26 Weeks (n=197, 201, 189, 78) | 1 | 0 | 0 | 0
  HDL-C, Low, 26 Weeks (n=127, 137, 129, 52) | 9 | 13 | 8 | 1
  HDL-C, High, 104 Weeks (n=206, 212, 199) | 2 | 1 | 2 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  HDL-C, Low, 104 Weeks (n=134, 143, 138) | 13 | 20 | 13 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  LDL-C, High, 26 Weeks (n=155, 163, 150, 61) | 15 | 11 | 19 | 7
  LDL-C, High, 104 Weeks (n=163, 170, 157) | 31 | 23 | 29 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  TG, High, 26 Weeks (n=163, 174, 156, 64) | 6 | 13 | 10 | 2
  TG, High, 104 Weeks (n=170, 183, 166) | 13 | 22 | 15 | NA — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.

22. Secondary Outcome: Change From Baseline in Pulse Rate at Dose Decision Point
Description: Sitting pulse rate was measured at the time that the dose decision was made (dose decision point). Change from baseline in pulse rate was 1 of the 4 measures included in the clinical utility index (CUI) used to evaluate the dose decision. The maximum duration of exposure to LY2189265, Sitagliptin, or Placebo (across all treatment arms) at the decision point was 27.4 weeks.
Time Frame: Baseline up to 27.4 weeks
Population: All participants randomized before the dose decision point who had evaluable sitting pulse rate data.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 14 | 30 | 23 | 9 | 20 | 22 | 17 | 35 | 33
beats per minute (bpm) | 6.63 (7.28) | 3.43 (10.14) | 2.39 (7.88) | 3.34 (9.88) | -1.63 (8.03) | 1.91 (6.18) | 1.05 (9.44) | -0.16 (8.07) | 1.81 (7.90)

23. Secondary Outcome: Change From Baseline in Blood Pressure at Dose Decision Point
Description: Sitting systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured at the dose decision point. Change from baseline in DBP was 1 of the 4 measures included in the clinical utility index (CUI) used to evaluate the dose decision. The maximum duration of exposure to LY2189265, Sitagliptin, or Placebo (across all treatment arms) at the time of the decision point was 27.4 weeks.
Time Frame: Baseline up to 27.4 weeks
Population: All participants randomized before the dose decision point who had evaluable sitting SBP and DBP data.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 14 | 30 | 23 | 9 | 20 | 22 | 17 | 35 | 33
millimeters of mercury (mmHg)
  Sitting SBP | -8.85 (12.92) | -4.63 (15.28) | -4.77 (11.37) | -2.00 (9.94) | -6.21 (19.13) | 0.40 (11.51) | 1.67 (10.18) | -2.16 (10.62) | -0.61 (14.75)
  Sitting DBP | -1.21 (7.47) | -1.17 (6.32) | -1.20 (4.67) | -0.08 (8.00) | -3.18 (10.13) | -0.75 (7.99) | 1.28 (4.06) | -1.11 (6.65) | -0.22 (7.94)

24. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Sitting and standing pulse rate were measured. Least squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as covariate.
Time Frame: Baseline, 26 weeks, 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable pulse data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
beats per minute (bpm)
  Sitting, 26 Weeks (n=271, 278, 283, 138) | 2.57 (0.47) | 1.90 (0.47) | -0.11 (0.46) | -0.22 (0.65)
  Sitting, 104 Weeks (n=197, 192, 191) | 2.28 (0.53) | 2.77 (0.54) | -0.78 (0.53) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Standing, 26 Weeks (n=271, 277, 281, 138) | 3.24 (0.52) | 2.00 (0.52) | -0.24 (0.51) | -0.17 (0.71)
  Standing, 104 Weeks (n=197, 192, 191) | 2.26 (0.63) | 2.50 (0.64) | -1.06 (0.63) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.

25. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Sitting and standing systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured. Least squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks, 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable SBP and DBP data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
millimeters of mercury (mmHg)
  Sitting SBP, 26 Weeks (n=271, 278, 283, 138) | -1.73 (0.67) | -1.40 (0.67) | -1.94 (0.66) | 1.12 (0.92)
  Sitting SBP, 104 Weeks (n=197, 192, 191) | -0.07 (0.81) | 1.28 (0.82) | 0.02 (0.82) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Sitting DBP, 26 Weeks (n=271, 278, 283, 138) | -0.43 (0.43) | -0.20 (0.43) | -1.06 (0.42) | 0.68 (0.58)
  Sitting DBP, 104 Weeks (n=197, 192, 191) | 0.38 (0.52) | 1.40 (0.52) | -0.36 (0.52) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Standing SBP, 26 Weeks (n=271, 277, 281, 138) | -1.53 (0.76) | -1.72 (0.76) | -2.54 (0.74) | 0.26 (1.04)
  Standing SBP, 104 Weeks (n=197, 192, 191) | -1.30 (0.92) | 0.17 (0.93) | -1.20 (0.92) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  Standing DBP, 26 Weeks (n=271, 277, 281, 138) | -0.11 (0.48) | 0.03 (0.48) | -1.36 (0.47) | -0.52 (0.66)
  Standing DBP, 104 Weeks (n=197, 192, 191) | -0.23 (0.57) | 0.36 (0.58) | -0.67 (0.58) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.

26. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters, Fridericia-corrected QT (QTcF) and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks, 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and comparator (Sitagliptin, Placebo/Sitagliptin) arms who had evaluable ECG data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks)
Number analyzed (Participants) | 304 | 302 | 315 | 177
milliseconds (msec)
  PR Interval, 26 Weeks (n=256, 261, 268, 132) | 2.94 (0.66) | 1.60 (0.66) | 0.42 (0.65) | 2.24 (0.89)
  PR Interval, 104 Weeks (n=168, 170, 167) | 4.59 (0.90) | 3.06 (0.90) | 3.19 (0.90) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.
  QTcF Interval, 26 Weeks (n=258, 262, 268, 132) | -3.86 (0.75) | -2.44 (0.75) | -1.31 (0.73) | 1.76 (1.02)
  QTcF Interval, 104 Weeks (n=169, 170, 168) | -2.71 (0.84) | -2.49 (0.84) | -0.02 (0.83) | NA (NA) — Placebo treatment lasted through 26 weeks. Thus, there are no data for this treatment arm at this time point.

27. Secondary Outcome: Participant-reported Outcomes, Impact of Weight on Quality of Life-Lite (IWQoL-Lite)
Description: The Impact of Weight on Quality of Life-Lite (IWQoL-Lite questionnaire) is an obesity-specific, 31-item questionnaire designed to measure the impact of weight on participants' quality of life. Items are scored on a 5-point numeric rating scale where 5 = "always true" and 1 = "never true". Items are summed into 6 scales (physical function [11 items], self-esteem [7 items], sexual life [4 items], public distress [5 items], work [4 items], and total score [31 items]) based on the average for the valid responses on that scale multiplied by the number of items on that scale (rounded to the nearest whole integer). Higher scores indicate lower levels of functioning (negative effects). Scores are linearly transformed to a 0 to 100 scale.
Time Frame: Baseline, 52 weeks, and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and active comparator (Sitagliptin) arms who had evaluable IWQoL-Lite data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 304 | 302 | 315
units on a scale
  Total Score, Baseline (n=285, 284, 300) | 83.41 (16.031) | 82.55 (16.952) | 83.97 (16.514)
  Total Score, 52 Weeks (n=237, 252, 247) | 86.92 (14.972) | 86.31 (14.673) | 86.25 (15.628)
  Total Score, 104 Weeks (n=190, 190, 185) | 88.08 (15.555) | 87.47 (15.183) | 86.93 (16.304)

28. Secondary Outcome: Participant-reported Outcomes, EQ-5D
Description: The EQ-5D questionnaire is a generic, multidimensional, health-related, quality-of-life instrument. It consists of 2 parts. The first part allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a three level scale of 1-3 (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the United Kingdom (UK) population-based algorithm. The possible values for the Index Score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension). The second part of the questionnaire consists of a 100-millimeter visual analog scale (VAS) on which the participants rated their perceived health state on that day from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, 52 weeks, and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and active comparator (Sitagliptin) arms who had evaluable EQ-5D data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 304 | 302 | 315
units on a scale
  EQ-5D, UK, Baseline (n=285, 281, 300) | 0.80 (0.222) | 0.82 (0.223) | 0.84 (0.216)
  EQ-5D, UK, 52 Weeks (n=237, 250, 244) | 0.83 (0.211) | 0.84 (0.208) | 0.85 (0.210)
  EQ-5D, UK, 104 Weeks (n=189, 190, 185) | 0.84 (0.203) | 0.86 (0.184) | 0.86 (0.198)
  VAS, Baseline (n=285, 284, 301) | 75.57 (15.798) | 75.35 (16.001) | 76.85 (15.363)
  VAS, 52 Weeks (n=238, 251, 245) | 78.93 (13.352) | 78.22 (13.839) | 78.79 (14.567)
  VAS, 104 Weeks (n=189, 190, 185) | 79.66 (13.820) | 78.52 (14.114) | 81.34 (13.708)

29. Secondary Outcome: Resource Utilization
Description: The number of visits to the emergency room (ER) is summarized cumulatively.
Time Frame: Baseline through 52 and 104 weeks
Population: All randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) and active comparator (Sitagliptin) arms.
Measure: Number; unit: events
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Sitagliptin
Number analyzed (Participants) | 304 | 302 | 315
events
  52 Weeks | NA — Data were not summarized cumulatively for this outcome measure. | NA — Data were not summarized cumulatively for this outcome measure. | NA — Data were not summarized cumulatively for this outcome measure.
  104 Weeks | NA — Data were not summarized cumulatively for this outcome measure. | NA — Data were not summarized cumulatively for this outcome measure. | NA — Data were not summarized cumulatively for this outcome measure.

30. Secondary Outcome: Pharmacokinetics of LY2189265: Area Under the Concentration-Time Curve
Description: Pharmacokinetic (PK) parameter estimates from LY2189265 concentration data were obtained using a 2-compartment population PK model with first order absorption. Area under the plasma-concentration curve from 0 to 168 hours, steady state (AUC0-168h, ss) of LY2189265 is summarized.
Time Frame: Baseline through 52 weeks
Population: Randomized participants in the selected (1.5 mg, 0.75 mg LY2189265) who had blood samples collected for PK assessments.
Measure: Mean (Standard Deviation); unit: nanograms times hours per milliliter
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265
Number analyzed (Participants) | 69 | 60
nanograms times hours per milliliter | 13378 (6100) | 7246 (3304)

31. Secondary Outcome: Antibodies to LY2189265
Description: The number of participants with postbaseline detection of treatment-emergent antidrug LY2189265 antibodies (ADA) is summarized.
Time Frame: Baseline through 104 weeks
Population: All randomized participants in the LY2189265 arms who had evaluable ADA data. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Number; unit: participants
Groups:
- LY2189265: LY2189265 (Dulaglutide): 3.0, 2.0, 1.5, 1.0, 0.75, 0.5, or 0.25 milligrams (mg), subcutaneous (SC), once weekly for up to 104 weeks.
  Placebo: tablet, administered orally, once daily for up to 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for up to 104 weeks
Arm/Group | LY2189265
Number analyzed (Participants) | 698
participants | 9

32. Other Pre Specified Outcome: Number of Participants With Adjudicated Pancreatitis at 104 Weeks
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 104 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Groups:
- Placebo/Sitagliptin (26 Weeks Through 104 Weeks): Placebo: solution, subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 26 weeks
  Sitagliptin: after 26 weeks, 100-milligrams (mg) tablet, administered orally, once daily for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks) | Placebo/Sitagliptin (26 Weeks Through 104 Weeks)
Number analyzed (Participants) | 15 | 30 | 304 | 10 | 302 | 25 | 24 | 315 | 177 | 177
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1

33. Other Pre Specified Outcome: Number of Participants With Adjudicated Cardiovascular Events at 104 Weeks
Description: Data on any new cardiovascular (CV) event was prospectively collected using a CV event electronic case report form. At prespecified visits, participants were asked about any new CV event. Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular AEs to be adjudicated include myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. The number of participants with adjudicated CV events is summarized cumulatively. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 104 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 26 Weeks) | Placebo/Sitagliptin (26 Weeks Through 104 Weeks)
Number analyzed (Participants) | 15 | 30 | 304 | 10 | 302 | 25 | 24 | 315 | 177 | 177
participants
  Participants With Any CV Event | 0 | 0 | 6 | 0 | 4 | 0 | 0 | 5 | 0 | 3
  Participants With a Fatal CV Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Participants With a Non-fatal CV Event | 0 | 0 | 6 | 0 | 4 | 0 | 0 | 4 | 0 | 2

ADVERSE EVENTS:
Groups:
- 0.75 mg LY2189265: LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 104 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally, for 104 weeks
- Placebo/Sitagliptin (Baseline Through 104 Weeks): Placebo: solution, subcutaneous (SC) injection, once weekly for 104 weeks
  Placebo: tablet, administered orally, once daily for 26 weeks
  Sitagliptin: after 26 weeks, 100-milligrams (mg) tablet, administered orally, once daily, for 78 weeks
  Metformin: at least 1500 milligrams per day (mg/day), administered orally for 104 weeks
Arm/Group | 3.0 mg LY2189265 | 2.0 mg LY2189265 | 1.5 mg LY2189265 | 1.0 mg LY2189265 | 0.75 mg LY2189265 | 0.5 mg LY2189265 | 0.25 mg LY2189265 | Sitagliptin | Placebo/Sitagliptin (Baseline Through 104 Weeks)
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/30 | 36/304 | 0/10 | 23/302 | 1/25 | 0/24 | 32/315 | 17/177
Other Adverse Events (participants affected / at risk) | 9/15 | 20/30 | 252/304 | 8/10 | 255/302 | 15/25 | 10/24 | 239/315 | 138/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 3.0 mg LY2189265 (N=15) | 2.0 mg LY2189265 (N=30) | 1.5 mg LY2189265 (N=304) | 1.0 mg LY2189265 (N=10) | 0.75 mg LY2189265 (N=302) | 0.5 mg LY2189265 (N=25) | 0.25 mg LY2189265 (N=24) | Sitagliptin (N=315) | Placebo/Sitagliptin (Baseline Through 104 Weeks) (N=177)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event resulted in death
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event resulted in death
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0/10 (0) | 0/22 (0) | 1/158 (1) | 0/7 (0) | 0/168 (0) | 0/12 (0) | 0/15 (0) | 0/164 (0) | 0/87 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0/10 (0) | 0/22 (0) | 1/158 (1) | 0/7 (0) | 0/168 (0) | 0/12 (0) | 0/15 (0) | 0/164 (0) | 0/87 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-secretory adenoma of pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5 (0) | 0/8 (0) | 0/146 (0) | 0/3 (0) | 0/134 (0) | 0/13 (0) | 0/9 (0) | 1/151 (1) | 0/90 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5 (0) | 0/8 (0) | 1/146 (1) | 0/3 (0) | 1/134 (1) | 0/13 (0) | 0/9 (0) | 0/151 (0) | 0/90 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/10 (0) | 0/22 (0) | 0/158 (0) | 0/7 (0) | 0/168 (0) | 0/12 (0) | 0/15 (0) | 1/164 (1) | 0/87 (0) — Event resulted in death
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/10 (0) | 0/22 (0) | 1/158 (1) | 0/7 (0) | 0/168 (0) | 0/12 (0) | 0/15 (0) | 0/164 (0) | 0/87 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Event resulted in death
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/10 (0) | 0/22 (0) | 0/158 (0) | 0/7 (0) | 0/168 (0) | 0/12 (0) | 0/15 (0) | 0/164 (0) | 1/87 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.0 mg LY2189265 (N=15) | 2.0 mg LY2189265 (N=30) | 1.5 mg LY2189265 (N=304) | 1.0 mg LY2189265 (N=10) | 0.75 mg LY2189265 (N=302) | 0.5 mg LY2189265 (N=25) | 0.25 mg LY2189265 (N=24) | Sitagliptin (N=315) | Placebo/Sitagliptin (Baseline Through 104 Weeks) (N=177)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3) | 10 (17) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 7 (7) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 13 (14) | 1 (1) | 15 (18) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 21 (26) | 0 (0) | 13 (24) | 1 (1) | 0 (0) | 11 (12) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 14 (15) | 0 (0) | 12 (13) | 1 (1) | 0 (0) | 9 (10) | 10 (12)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 14 (14) | 0 (0) | 16 (22) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 50 (74) | 1 (1) | 36 (53) | 4 (5) | 2 (2) | 18 (30) | 15 (23)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 18 (25) | 1 (1) | 19 (23) | 3 (4) | 1 (1) | 16 (17) | 4 (4)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (9) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 11 (12) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 9 (9) | 7 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 7 (8) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 7 (7) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (6) | 53 (98) | 4 (5) | 44 (62) | 3 (6) | 2 (3) | 22 (27) | 9 (15)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (6) | 41 (62) | 2 (2) | 25 (43) | 1 (1) | 1 (2) | 11 (11) | 3 (3)
Asthenia (General disorders) | 0 (0) | 2 (3) | 7 (8) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 13 (15) | 1 (1) | 9 (9) | 0 (0) | 2 (2) | 11 (11) | 6 (6)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 12 (12) | 0 (0) | 7 (10) | 1 (1) | 0 (0) | 6 (6) | 7 (8)
Influenza (Infections and infestations) | 0 (0) | 1 (2) | 16 (19) | 0 (0) | 18 (22) | 0 (0) | 0 (0) | 14 (15) | 5 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 43 (64) | 0 (0) | 48 (96) | 1 (1) | 0 (0) | 47 (72) | 25 (44)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 15 (22) | 0 (0) | 10 (14) | 2 (2) | 0 (0) | 7 (7) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 22 (34) | 0 (0) | 22 (30) | 1 (1) | 0 (0) | 21 (24) | 7 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 21 (26) | 0 (0) | 21 (25) | 1 (1) | 1 (1) | 19 (22) | 14 (21)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 6 (11) | 1 (1) | 5 (9) | 1 (1) | 0 (0) | 6 (8) | 1 (1)
Blood calcitonin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 11 (14) | 0 (0) | 13 (21) | 2 (2) | 1 (1) | 15 (16) | 5 (9)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 29 (31) | 1 (1) | 17 (23) | 2 (2) | 1 (1) | 11 (11) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 30 (30) | 0 (0) | 38 (38) | 0 (0) | 0 (0) | 49 (49) | 28 (28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 15 (19) | 0 (0) | 19 (22) | 0 (0) | 0 (0) | 14 (16) | 7 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 21 (28) | 0 (0) | 28 (32) | 2 (2) | 0 (0) | 19 (24) | 9 (9)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 7 (8) | 0 (0) | 18 (20) | 0 (0) | 0 (0) | 14 (20) | 6 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 29 (53) | 0 (0) | 27 (76) | 1 (1) | 1 (3) | 26 (33) | 12 (17)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 7 (10) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 7 (8) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 19 (24) | 0 (0) | 11 (12) | 0 (0) | 0 (0) | 17 (26) | 6 (7)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days